CLINICAL TRIAL: NCT06899126
Title: A Phase 3, Multicenter, Randomized, Open-label Trial of Trastuzumab Deruxtecan in Combination With Pembrolizumab Versus Platinum-based Chemotherapy in Combination With Pembrolizumab, as First-line Therapy in Participants With Locally Advanced Unresectable or Metastatic HER2 Overexpressing and PD-L1 TPS <50% Non-squamous Non-small Cell Lung Cancer (DESTINY-Lung06)
Brief Title: Study of Trastuzumab Deruxtecan, Pembrolizumab, and Platinum-based Chemotherapy in First-line HER2 Overexpressing Non-small Cell Lung Cancer
Acronym: DESTINY-Lung06
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS8201-793; 2024-515658-26-00 (EU CTIS Number); KEYNOTE-G23 (Other: Merck Sharp & Dohme LLC); MK-3475-G23 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2025-03-21; First posted 2025-03-27 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: DESTINY; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — trastuzumab deruxtecan; pembrolizumab; Pemetrexed; Drug Therapy

STUDY DESIGN:
Masking Description: This is an open-label study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: T-DXd (Experimental): Participants will receive T-DXd plus pembrolizumab
  Interventions: Drug: Trastuzumab Deruxtecan; Drug: pembrolizumab
- Arm B: Pemetrexed + Chemotherapy + Pembrolizumab (Active Comparator): Participants will receive Pemetrexed plus platinum chemotherapy (cisplatin or carboplatin) plus pembrolizumab
  Interventions: Drug: pembrolizumab; Drug: Pemetrexed; Drug: Chemotherapy

INTERVENTIONS:
Drug: Trastuzumab Deruxtecan — T-DXd will be administered at a dose of 5.4 mg/kg intravenously (IV) every 3 weeks (Q3W)
  Other Names: T-DXd; ENHERTU®; DS-8201a
  Arms: Arm A: T-DXd
Drug: pembrolizumab — pembrolizumab will be administered at a dose of 200 mg IV Q3W
  Other Names: KEYTRUDA®
Drug: Pemetrexed — Pemetrexed will be administered at a dose of 500 mg/m2 IV Q3W
  Arms: Arm B: Pemetrexed + Chemotherapy + Pembrolizumab
Drug: Chemotherapy — One of the following two will be administered in Arm B:
  Cisplatin at a dose of 75 mg/m2 IV or carboplatin AUC at a dose of 5 mg/mL/min IV
  Arms: Arm B: Pemetrexed + Chemotherapy + Pembrolizumab

SUMMARY:
This clinical trial is designed to assess the efficacy and safety of trastuzumab deruxtecan (T-DXd; Enhertu®) in combination with pembrolizumab versus platinum-based chemotherapy in combination with pembrolizumab in participants with no prior therapy for locally advanced unresectable or metastatic non-squamous NSCLC, whose tumors have HER2-overexpressing and PD-L1 TPS <50% without known AGA that have locally available therapies targeting their AGAs in first-line advanced/metastatic setting.

ELIGIBILITY:
Inclusion Criteria:

1. Sign and date the Tissue Screening ICF, prior to any Tissue Screening procedure. Sign and date the Main ICF, prior to the start of any trial-specific qualification procedures.

   Sign and date the Optional PGx ICF (included in the Main Screening ICF) prior to any PGx procedure, and the Pregnant Partner ICF, if applicable.
2. Adults ≥18 years of age on the day of signing the ICF. Follow local regulatory requirements if the legal age of consent for trial participation is >18 years old.
3. Histologically documented non-squamous locally advanced unresectable or metastatic

   NSCLC and meets all of the following criteria:

   Has Stage IV NSCLC disease or Stage IIIB or IIIC disease but is not a candidate for surgical resection or definitive chemoradiation at the time of randomization (based on the American Joint Committee on Cancer, Eighth Edition). Has no known AGAs (based on existing test result of local test) that have locally available therapies targeting their AGAs in the first-line advanced/metastatic setting. Has no known HER2 mutation based on existing test results (if approved or validated local test is available). Note: Participants with mixed histology are eligible if adenocarcinoma is the predominant histology. Mixed tumors will be classified based on the predominant cell type.
4. Has not been treated with systemic anticancer therapy for advanced or metastatic non-squamous NSCLC. Participants who received adjuvant or neoadjuvant therapy other than those listed below, including ICI (ie, anti-PD-1/PD-L1) or a platinum-based regimen, are eligible if the last dose of adjuvant/neoadjuvant therapy was given at least 6 months before the date of the first trial dose and should not have progressed on or within 6 months of the last dose date of adjuvant/neoadjuvant therapy.

   1. Any agent, including an ADC, containing a chemotherapeutic agent targeting topoisomerase I.
   2. HER2-targeted antibody-based anticancer therapy.
5. Has adequate tumor tissue sample (not previously irradiated) available for assessment of HER2 and PD-L1 expression by central or Sponsor-specified laboratory. A new biopsy is required if the participant's most recent archival tumor tissue sample cannot be supplied.

Details pertaining to tumor tissue submission can be found in the Trial Laboratory Manual.

Exclusion Criteria:

1. Has a medical history of MI within 6 months before randomization/enrollment or symptomatic CHF (NYHA Class II to Class IV). Participants with troponin levels above the ULN at Screening (as defined by the manufacturer) and without any MI-related symptoms should have a cardiologic consultation during the Screening Period to rule out MI.
2. Has a QTc prolongation to >480 ms based on the average of the Screening triplicate 12- lead ECG.
3. Has a history of (non-infectious) ILD/pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at Screening.
4. Has lung-specific, intercurrent, clinically significant illnesses including, but not limited to, any underlying pulmonary disorder (eg, pulmonary emboli within 3 months of the trial randomization, severe asthma, severe COPD, restrictive lung disease, pleural effusion, etc.).
5. Had a prior complete pneumonectomy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2025-10-24 (Actual); Primary Completion 2030-03-05 (Estimated); Study Completion 2032-07-05 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival by Blinded Independent Central Review | From date of randomization to the date of radiographic disease progression or death due to any cause, up to 54 months
  PFS is defined as the time interval from the date of randomization to the date of radiographic disease progression or death due to any cause. Tumor response will be determined by BICR assessment of tumor scans using RECIST v1.1.

SECONDARY OUTCOMES:
Overall Survival | From date of randomization to the date of death due to any cause, up to 85 months
  OS is defined as the time interval from the date of randomization to the date of death due to any cause.

CONTACTS AND LOCATIONS:
Locations (100):
- United States (18):
  - Alaska Oncology & Hematology, LLC, Anchorage, Alaska
  - Orange Coast Memorial Medical Center Fountain Valley, Fountain Valley, California
  - California Research Institute, Los Angeles, California
  - Los Angeles Cancer Network (LACN), Los Angeles, California
  - Providence Medical Foundation, Santa Rosa, California
  - Bay Pines VA Healthcare System, Bay Pines, Florida
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mid-Florida Hematology & Oncology Centers, P.A., Orange City, Florida
  - BRCR Global Plantation, Plantation, Florida
  - Hope and Healing Cancer Services, Hinsdale, Illinois
  - Logan Health Research, Kalispell, Montana
  - Clinical Research Alliance, Westbury, New York
  - FirstHealth Cancer Center, Pinehurst, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - St. Charles Health System, Bend, Oregon
  - University of Texas M. D. Anderson Cancer Center, Houston, Texas
  - Lumi Research, Kingwood, Texas
  - Summit Cancer Treatment Center, Spokane, Washington
- Argentina (4):
  - CINME - Centro De Investigaciones Metabolicas, Buenos Aires
  - Instituto Argentino de Diagnostico y Tratamiento, Buenos Aires
  - Instituto de Investigaciones Metabolicas (IDIM), Buenos Aires
  - Instituto Medico de la Fundacion Estudios Clinicos, Rosario
- CHU Helora-Hospital de Mons, Mons, Belgium
- Brazil (13):
  - Hospital de Cancer de Barretos - Fundacao Pio XII, Barretos
  - Centro de Pesquisas Clinica Reichow, Blumenau
  - CIONC-Centro Integrado de Oncologia de Curitiba, Curitiba
  - CRIO - Centro Regional Integrado de Oncologia, Fortaleza
  - Liga Norte-Rio-Grandense Contra o Câncer, Natal
  - Hospital Ernesto Dornelles, Porto Alegre
  - Hospital São Lucas da PUCRS, Porto Alegre
  - Centro de Tratamento Oncologico (CTO), Ribeirão Preto
  - Hospital das Clínicas FMRP-USP, Ribeirão Preto
  - Obras Sociais Irmã Dulce - Hospital Santo Antônio, Salvador
  - CEPHO - Centro de Estudos e Pesquisas de Hematologia e Oncologia, Santo André
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto, Sao Jose Rio Preto
  - Centro Paulista de Oncologia S A, Vila Olímpia
- China (23):
  - China-Japan Friendship hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Sichuan Cancer Hospital, Chengdu
  - West China Hospital, Sichuan University, Chengdu
  - Chongqing University Cancer Hospital, Chongqing
  - Nanfang Hospital of Southern Medical University, Guangzhou
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - The Second Hospital of Anhui Medical University, Hefei
  - Hong Kong Integrated Oncology Centre, Hong Kong
  - Cancer Hospital of Shandong First Medical University, Jinan
  - Hong Kong United Oncology Centre, Jordan
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - The Second People's Hospital of Neijiang, Neijiang
  - Shanghai East Hospital, Shanghai
  - Liaoning Cancer Hospital & Institute, Shenyang
  - Shanxi Provincial Cancer Hospital, Taiyuan
  - Tianjin Medical University General Hospital, Tianjin
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Xiangyang Central Hospital, Xiangyang
- Hopital Albert Calmette - CHU Lille, Lille, France
- Japan (19):
  - Saitama Medical University International Medical Center, Hidaka-shi
  - Kansai Medical University Hospital, Hirakata-shi
  - Hirosaki University Hospital, Hirosaki-shi
  - St. Marianna University Hospital, Kawasaki-shi
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi
  - Saiseikai Kumamoto Hospital, Kumamoto
  - Kurume University Hospital, Kurume-shi
  - Matsusaka Municipal Hospital, Matsusaka-shi
  - NHO Okayama Medical Center, Okayama
  - Osaka City General Hospital, Osaka
  - Osaka International Cancer Institute, Osaka
  - NHO Kinki-Chuo Chest Medical Center, Sakaishi
  - Keijinkai Teine Keijinkai Hospital, Sapporo
  - Tokyo Medical University Hospital, Shinjuku-ku
  - Shizuoka Cancer Center, Sunto-gun
  - Fujita Health University Hospital, Toyoake-shi
  - Wakayama Medical University Hospital, Wakayama
  - Kanagawa Cancer Center, Yokohama
  - Tottori University Hospital, Yonago-shi
- Malaysia (3):
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Hospital Tengku Ampuan Afzan, Kuantan
  - Beacon Hospital Sdn Bhd, Petaling Jaya
- Unidade Local de Saude de Santa Maria, E.P.E. - Hospital Pulido Valente, Lisbon, Portugal
- South Korea (8):
  - National Cancer Center, Goyang-si
  - Gyeongsang National University Hospital, Jinju
  - CHA Bundang Medical Center, CHA University, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - The Catholic University of Korea, St. Vincent's Hospital, Suwon
- Taiwan (8):
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - Taichung Veterans General Hospital, Taichung
  - Chi Mei Hospital, Liouying, Tainan
  - National Cheng Kung University Hospital, Tainan
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Chang Gung Memorial Hospital,Linkou, Taoyuan
- Charing Cross Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) on completed studies and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Completed studies that has reached a global end or completion with all data set collected and analyzed, and for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents on completed clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/